CLINICAL TRIAL: NCT05968924
Title: Improving DFU Outcomes: Early Detection of Foot Ulcers Using Novel Technology
Acronym: DFUMAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: Podimetrics, Inc. (Industry); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2023-14915; P30DK111022 (NIH)
Record Dates: First submitted 2023-07-20; First posted 2023-08-01 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Diabetic Foot Ulcer
Keywords: Diabetes; Foot Ulcer; Prevention; Innovation
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus; Foot Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- High risk Diabetic Foot Ulcer (DFU) (Experimental): Podimetrics smart map
  Interventions: Device: Podimetrics SmartMat

INTERVENTIONS:
Device: Podimetrics SmartMat — Participants receive training for stepping on SmartMat each day for 6 months. Monthly phone calls will be conducted to assess foot health and mat.

SUMMARY:
The investigator team will study the adherence of the participant cohort to a non significant risk device over a six month period. The device is a foot mat, which can detect changes in foot temperature that may predict foot ulceration in patients with diabetes mellitus. This mat, the Podimetrics Smart Mat, is FDA cleared.

DETAILED DESCRIPTION:
Innovations toward the prevention of diabetic foot ulcer (DFU) are needed. Early detection of changes in the foot that predict the development of DFU could allow timely intervention to prevent the limb damage that occurs with advanced DFU.

Studies have demonstrated that increased temperature in the foot presage the development of DFU. Temperature changes can accurately be detected by home monitoring devices and predict impending ulceration. Here the study team will test the uptake of novel foot temperature monitoring technology for a future intervention study to determine if a home monitoring device could prevent the occurrence of severe DFU for patients at Montefiore Medical Center (MMC).

The investigator team will conduct a longitudinal study to determine the adherence to an FDA cleared device, Podimetrics, which has been tested in other populations and shown to 1) decrease the risk of severe DFU, and 2) decrease the utilization of health care resources in high risk patients with a history of DFU.

For this study, the study team will identify and enroll patients who are at high risk for DFU. These participants will be identified from the electronic medical record (EMR) and have case report form filled out.

After providing informed consent, study participants will receive the foot mat and obtain training remotely from Podimetrics, which provides a standardized training program.

Participants briefly stand on the mat daily (20 seconds), and the temperature data is automatically sent for analysis to Podimetrics to interpret the information. The participants will be evaluated over a six-month period to measure:

1. Daily use of the technology
2. Secondary outcomes: occurrence of DFU and use of health care resources.

Study participants will be contacted every month by the Einstein investigators to assess foot health. Study participants will be instructed to contact the study team during the study period to inquire if development of any changes in the foot such as the diagnosis of DFU, or if a foot cast is required for offloading, or if participants have any concerns about their feet.

ELIGIBILITY:
Inclusion Criteria:

1. Type 1 or Type 2 diabetes mellitus
2. Prior treatment of DFU within 24 months
3. Subject had at least one outpatient follow up with a provider after treatment for DFU
4. No active ulcer at time of enrollment
5. Male or female, aged 18-75 yrs
6. Presence of Neuropathy
7. Ambulatory
8. Provision of signed and dated informed consent form
9. Stated willingness to adhere with all study procedures and availability to participate for the duration of the study

Exclusion Criteria:

1. Active diabetic foot ulcer (DFU)
2. Unable to comply with study requirements
3. Prior above-knee amputation (AKA) or below-knee amputation (BKA)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-07-03 (Actual); Primary Completion 2025-04-03 (Actual); Study Completion 2025-04-03 (Actual)

PRIMARY OUTCOMES:
Adherence to use of SmartMat | Six months
  Participant adherence to use of SmartMat will be quantified by automated data collection. % of daily use over 6 months will be summarized and reported.

SECONDARY OUTCOMES:
Use of health care facilities | Up to six months
  Enumerate total number of health care visits over the course of the study. This will include patient visits to the Emergency Room (ER), podiatrist, internist, walk in clinic, and other health care facilities and will be be based on subject self-reporting of visits.
Occurrence of Diabetic Foot Ulcer (DFU) | Up to six months
  The number of participants who develop DFU during the course of the study will be summarized and reported.

CONTACTS AND LOCATIONS:
Overall Officials: Johanna Daily, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Armstrong DG, Holtz-Neiderer K, Wendel C, Mohler MJ, Kimbriel HR, Lavery LA. Skin temperature monitoring reduces the risk for diabetic foot ulceration in high-risk patients. Am J Med. 2007 Dec;120(12):1042-6. doi: 10.1016/j.amjmed.2007.06.028. PMID 18060924
- [Background] Crocker RM, Palmer KNB, Marrero DG, Tan TW. Patient perspectives on the physical, psycho-social, and financial impacts of diabetic foot ulceration and amputation. J Diabetes Complications. 2021 Aug;35(8):107960. doi: 10.1016/j.jdiacomp.2021.107960. Epub 2021 May 23. PMID 34059410
- [Background] Hoban C, Sareen J, Henriksen CA, Kuzyk L, Embil JM, Trepman E. Mental health issues associated with foot complications of diabetes mellitus. Foot Ankle Surg. 2015 Mar;21(1):49-55. doi: 10.1016/j.fas.2014.09.007. Epub 2014 Sep 22. PMID 25682407
- [Background] Isaac AL, Swartz TD, Miller ML, Short DJ, Wilson EA, Chaffo JL, Watson ES, Hu H, Petersen BJ, Bloom JD, Neff NJ, Linders DR, Salgado SJ, Locke JL, Horberg MA. Lower resource utilization for patients with healed diabetic foot ulcers during participation in a prevention program with foot temperature monitoring. BMJ Open Diabetes Res Care. 2020 Oct;8(1):e001440. doi: 10.1136/bmjdrc-2020-001440. PMID 33055233
- [Background] Lavery LA, Higgins KR, Lanctot DR, Constantinides GP, Zamorano RG, Armstrong DG, Athanasiou KA, Agrawal CM. Home monitoring of foot skin temperatures to prevent ulceration. Diabetes Care. 2004 Nov;27(11):2642-7. doi: 10.2337/diacare.27.11.2642. PMID 15504999
- [Background] Margolis DJ, Malay DS, Hoffstad OJ, Leonard CE, MaCurdy T, de Nava KL, Tan Y, Molina T, Siegel KL. Incidence of diabetic foot ulcer and lower extremity amputation among Medicare beneficiaries, 2006 to 2008. 2011 Feb 17. In: Data Points Publication Series [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2011-. Data Points #2. Available from http://www.ncbi.nlm.nih.gov/books/NBK65149/ PMID 22049565
- [Background] Rothenberg GM, Page J, Stuck R, Spencer C, Kaplan L, Gordon I. Remote Temperature Monitoring of the Diabetic Foot: From Research to Practice. Fed Pract. 2020 Mar;37(3):114-124. PMID 32317847
- [Background] Skafjeld A, Iversen MM, Holme I, Ribu L, Hvaal K, Kilhovd BK. A pilot study testing the feasibility of skin temperature monitoring to reduce recurrent foot ulcers in patients with diabetes--a randomized controlled trial. BMC Endocr Disord. 2015 Oct 9;15:55. doi: 10.1186/s12902-015-0054-x. PMID 26452544